CLINICAL TRIAL: NCT02863744
Title: Estimation of MMP-8 Levels in GCF and Serum and Its Correlation With Wound Healing and Clinical Outcomes After Coronally Advanced Flap and Subepithelial Connective Tissue Graft for Root Coverage in Recession Defects: A CLINICO-BIOCHEMICAL STUDY
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: 6 month follow up for the patients in progress
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-D012-54506
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Wound Healing
Keywords: mmp-8; early stages of wound healing; wound healing marker

ARMS (1):
- CAF+SCTG (Experimental)
  Interventions: Procedure: coronally advanced flap with subepithelial connective tissue graft

INTERVENTIONS:
Procedure: coronally advanced flap with subepithelial connective tissue graft — * Under local anesthesia 2% lignocaine hydrochloride using a No. 15 BP (Bard Parker) blade full thickness flap will be elevated till the MGJ (mucogingival junction) using a small periosteal elevator and a partial-thickness flap will be raised beyond the mucogingival junction to allow a passive coronal displacement of the flap completely covering the CEJ without tension.
  * The donor site consisting of 2 mm thick palatal connective tissue graft will be harvested from the premolar to the first molar area using the 'trap door' technique.14 The connective tissue graft will be secured in position with 4-0 absorbable sutures in recipient sites.
  The flaps will be stabilized with sling suture in a coronal position, followed by interrupted suture on releasing incisions in an apico-coronal direction using 4-0 absorbable sutures.

SUMMARY:
Assessment of wound healing progression after surgery is important. Currently blunt surrogate markers such as probing is used. Limitation of these markers is that it represents the history of healing and not the ongoing activity. As hallmark of healing is collagen remodeling, it is of interest to study the cytokine profile that relates to wound healing. Such knowledge may potentially lead to new diagnostic strategies to study wound healing in a better way reflecting the healing phenotype. Understanding wound healing at molecular level provides an in depth basis to develop treatment strategies that can prevent delayed healing.2 As recommended by Consensus Report of 10th European workshop on periodontology that, there is a need for more studies at cellular level to identify cytokine, chemokine, and intracellular signaling networks for better regenerative approaches10, the present clinical trial was designed.

On account of a considerable lacunae in this area of periodontal research, this study is planned to assess the MMP-8 levels during the post-op healing following CAF+SCTG surgery for recession coverage and to better identify the mechanism involved in wound healing. This information can be used to prevent the normal surgical wound from altered healing experience.

DETAILED DESCRIPTION:
NEED FOR THE STUDY:

Coronally advanced flap with Subepithelial Connective Tissue Graft (CAF+SCTG) technique has proven to be one of the most successful modalities for root coverage.1 The success of any surgical procedure is dependent on wound healing.

Wound healing after surgical procedure is complex and highly orchestrated event that includes hemostatic phase, inflammatory phase, phase of new tissue formation and the final remodelling phase leaving behind collagen rich extracellular matrix (ECM) and a dense and stable tissue.2 During wound healing clot provides a foundation for the future ECM. ECM plays a vital role to prompt cellular migration, adhesion, wound contraction and epithelialization. This crucial role of ECM is maintained by a group of enzymes collectively known as Matrix Metalloproteinases (MMPs). MMPs plays a central role in wound healing.3,4 Failure of regulation of these MMPs has been correlated with faulty wound healing.3,4 MMPs (i.e. collagenases, gelatinases, matrilysins, stromelysins, and membrane type MMPs) are family of zinc dependent endopeptidases capable of cleaving extracellular matrix (ECM) in healing wounds.3 MMP-8 are primarly produced by neutrophils and are also produced by other cells such as oral epithelial cells, plasma cells and fibroblasts.7 MMP-8 is expressed during the myelocytic stage of development of PMN (Polymorphonuclear cell) precursors in the bone marrow29 and is stored as latent enzyme (pro-mmp-8) within the specific granules of PMN.30 Pro-MMP-8 is rapidly released from activated PMN undergoing degranulation31 and then is activated via cysteine switch mechanism to yield the active form of enzyme.29 MMP-8 (polymorphonuclear collagenase5) cleaves the triple helix of fibrillar collagen and has affinity for type I collagen and type III collagen5 that is abundantly found in connective tissue of gingiva. MMP-8 degrades gelatin type VII, VIII and X collagen.5 MMP-8 has been implicated to be important for acute wound healing.6 Assessment of wound healing progression after surgery is important. Currently blunt surrogate markers such as probing is used. Limitation of these markers is that it represents the history of healing and not the ongoing activity. As hallmark of healing is collagen remodeling, it is of interest to study the cytokine profile that relates to wound healing. Such knowledge may potentially lead to new diagnostic strategies to study wound healing in a better way reflecting the healing phenotype.

The function of collagenase during normal wound healing after periodontal surgery has been relatively ill-defined due to lack of studies in this area.10 Most of the research has concentrated on the characterisation of MMP-8 during pathogenesis of periodontal disease8 and the changes in MMP-8 level after periodontal treatment.

Nwomeh et al studied MMP-8 from dermal wound healing by collecting wound exudate from occlusive bandage. He noted that MMP-8 peaked at day 4 and persisted for about a week. MMP-8 over expression leads to faulty healing.5 Chronic wounds have 30 times greater MMPs than acute wounds. Inhibiting excessive protease expression in these wounds may allow a prospective wound healing treatment.5 Very less is known about the cellular aspects of soft tissue healing in the oral mucosa. The assumption that oral healing is similar to dermal wounds might provoke confusion, as there are certain subtle difference like reduced scar formation in the dermal wounds2, role of IL-1 in oral wounds and absence of IL-1 in dermal wounds11, faster healing in oral wounds, presence of saliva that aids in healing etc. Overall it is still a matter of speculation and ambiguity about the differences in the unique healing pattern of oral wounds.

Understanding wound healing at molecular level provides an in depth basis to develop treatment strategies that can prevent delayed healing.2 As recommended by Consensus Report of 10th European workshop on periodontology that, there is a need for more studies at cellular level to identify cytokine, chemokine, and intracellular signaling networks for better regenerative approaches10, the present clinical trial was designed.

On account of a considerable lacunae in this area of periodontal research, this study is planned to assess the MMP-8 levels during the post-op healing following CAF+SCTG surgery for recession coverage and to better identify the mechanism involved in wound healing. This information can be used to prevent the normal surgical wound from altered healing experience.

6.2 REVIEW OF LITERATURE: Sanctis et al. (2011) conducted a study to determine the use of connective tissue graft (CTG) in root coverage. The results proved CAF in association with SCTG is a valid approach in the treatment of recession defects Nwomeh et al. (1999) assessed the sources of collagenases (MMP-8, MMP-1) and their activity in normal healing wounds and chronic non healing ulcers. The results showed MMP-8 is predominant collagenase present in normal healing wounds and chronic non healing ulcers had increased level of MMP-1,8 and decreased levels of TIMP-1 Armstrong et al (2002) reviewed the key role of MMP-8 in wound healing as predominant collagenase. He elaborated the expressions of peak levels of MMP-8 at day 4 and 7 during normal wound healing.

Hammerle et al (2014) in a consensus report that reviewed the biological processes of soft tissue wound healing in oral cavity, found that oral soft tissue healing at teeth, implants and edentulous ridge follows the same phase as skin wound healing and human histological data are limited.

Sorsa et al (2010) compared four methods for gingival crevicular fluid matrix metalloproteinase (MMP-8) detection i.e., Immunofluorometeric assay, Dip stick test, dentoAnalyser immunoblot assay and ELISA kit in their study and concluded that all the assays are comparable and dentoAnalyser is among first quantitative MMP-8 chair side testing devices in periodontal and peri implant diagnostics and research.

Fernandez et al ( 2007 ) conducted a study to investigate the role of MMP_8 in cutaneous wound healing healing. They observed significant delay in wound closure in MMP-8 -/- mice and an altered inflammatory response in their wounds. They indicated that MMP-8 participates in wound repair by resolution of inflammation and open the possibility to develop new strategies for treating wound healing defects.

Mohd H et al (1999)19 assessed the levels of MMP-8 and MMP-3 during early healing phase following a guided tissue regeneration procedure by assessing GCF (Gingival Crevicular Fluid) samples for quantification of MMP-8 and MMP-3. They found that presence of the membrane appeared to increase the levels of MMP-3 and -8 and relate to the resorption of the bioresorbable membrane by host systems.

Dickinson et al (2013) studied the early events in periodontal regeneration in the canine supraalveolar periodontal defect model by using histologic and immunological techniques and concluded that activation of cellular regenerative events in periodontal wound regeneration is rapid, the general frame work of tissue formation ( bone, periodontal ligament, and Connective tissue) is broadly outlined within 14 days.

Shaw et al (2009) reviewed wound repair at a glance and described the complex process of wound repair. He emphasized that the remodeling of extracellular matrix is accomplished by a delicate balance of MMPs.

Teles et al (2010) measured the levels of GCF biomarkers and subgingival bacterial species in periodontally healthy and periodontitis subjects. He concluded that clinically healthy sites from periodontitis subjects present higher levels of GCF biomarkers and periodontal pathogens than sites from healthy subjects.

6.3 Objective of the study: The primary objective of this study is to evaluate the effect and impact of CAF+SCTG for root coverage in Millers class I and II gingival recession sites on the MMP-8 levels in GCF and serum.

The secondary objective is to test the utility of base line MMP-8 level in predicting categorically assessed treatment outcomes and correlate it with early wound healing pattern following CAF+SCTG for root coverage.

MATERIALS AND METHODS:

7.1 Source of data:

Patients visiting the outpatient Department of Periodontology, Krishnadevaraya College of Dental Sciences and Hospital and satisfying the inclusion and exclusion criteria will be screened and selected for the study.

The experimental design will be consisting of a total 15-20 sites who will be recruited for the study as per the inclusion and exclusion criteria. The patients will be informed about the surgical procedure and materials used for the study and an informed consent will be obtained from the patients.

7.2 Method of collection of data:

Sample size:

This prospective study will be a single blind comparative clinical control trial with 15-20 patients having Miller's class I and II recession defects in the maxillary anterior arch.

Sampling technique

* After screening examinations in the initial phase, each subject will receive a session of oral hygiene instructions, scaling and root planning with ultrasonic scalers and manual curettes.
* Surgical treatment of recession defect will not be scheduled until the patient can demonstrate an adequate standard of supragingival plaque control (plaque score <20% O Leary 1972). The below mentioned clinical parameters will be recorded to the nearest millimeter using a UNC-15-probe (University of North Carolina -15 periodontal probe -Hu Friedy, Chicago, IL, USA) and measuring occlusal stents for positioning measuring probes will be fabricated with cold-cured acrylic resin on a cast model obtained from an alginate impression. It will be constructed so that it covers the occlusal surfaces of the tooth being treated and the occlusal surfaces of at least one tooth in mesial and distal directions. It will also be extended apically on the buccal and lingual surfaces to cover the coronal third of the teeth. Three grooves will be marked on the stent at mesio-buccal, mid-buccal and disto-buccal sites as the reference points15 so that post surgical measurement will be made at the same position and angulation as those made before surgery ie baseline measurements then after 6 months.
* The GCF sample will be collected from gingival sulcus of the tooth indicated for root coverage procedure (negative control) and from another tooth wth clinically healthy gingiva (positive control). The samples will be collected at baseline and at subsequent post surgical followup (fourth day, seventh day and 6 months).

Clinical measurements:

The following clinical measurement will be recorded at baseline and after 6 months.

1. Gingival Recession depth (GRD), measured as the distance between the CEJ and gingival margin.17
2. Gingival Recession Width (GRW), measured as the distance between the mesial gingival margin and distal gingival margin.17
3. Probing Depth (PD), measured as the distance from gingival margin to the base of gingival sulcus.17
4. Clinical Attachment Level (CAL), measurement from the CEJ ( Cementoenamel junction) to the base of the gingival sulcus.17
5. Apico coronal width of keratinised tissue (KTW) measured as the distance from mucogingival junction to the gingival margin.17
6. Wound Healing indices (WHI) will be assessed on 4th and 7th day ( Lien-Hui Huang, 2005)
7. Plaque Index (Sillness and Loe, 1964)
8. Gingival Index (Loe and Sillness, 1963)
9. Gingival Bleeding Index (Ainamo and Bay, 1975)

SURGICAL PROCEDURE:

* Before starting the surgery, root surfaces near to buccal attachment loss will be instrumented with mini-five Gracey Currettes and the mechanical treatment will be terminated when smooth and hard root surfaces will be obtained.16
* Under local anesthesia 2% lignocaine hydrochloride (Ligox 2%, Indoco Remedies Ltd, Goa, India) using a No. 15 BP (Bard Parker) blade, a submarginal incision will be made at the buccal aspect of the treated tooth and extended 3 mm horizontally in the mesial and distal interdental gingiva. An intrasulcular incision will be made at the buccal aspect of the involved tooth. Two oblique, divergent releasing incisions will be followed, extending beyond the mucogingival junction.
* A full thickness flap will be elevated till the MGJ (mucogingival junction) using a small periosteal elevator. Subsequently, a partial-thickness flap will be raised beyond the mucogingival junction to allow a passive coronal displacement of the flap completely covering the CEJ without tension.16
* Root planning will be done using a sharp curette.The papillae adjacent to the treated tooth will be de-epithelialized to create a bleeding surface for a recipient bed, where SCTG will be placed.
* The donor site consisting of 2 mm thick palatal connective tissue graft will be harvested from the premolar to the first molar area using the 'trap door' technique.14 The connective tissue graft will be secured in position with 4-0 absorbable sutures in recipient sites.
* The flaps will be stabilized with sling suture in a coronal position, followed by interrupted suture on releasing incisions in an apico-coronal direction using 4-0 absorbable sutures.14
* The surgical sites will be protected with a non eugenol periodontal dressing. Post operative instructions will consist of 0.2% chlorhexidine mouth rinse 3 times daily for 3 weeks and Ibuprofen 600 mg for pain control for three days. 33
* Sutures will be removed 7 days after surgery and after this patients will be reinstructed in mechanical cleaning of treated teeth with use of soft toothbrush.33
* Recall and reinforcement of oral hygiene instructions will be done every 2 months.

Gingival crevicular fluid (GCF) sampling and ELISA:

* The subjects will be seated comfortably in an upright position on the dental chair, and the selected site will be well illuminated.
* GCF samples will be collected after plaque index but before any other clinical recordings which would cause tissue irritation and blood contamination of sample.19 During the 4th and 7th day post surgical follow up ,the periodontal dressing will be gently removed and GCF samples will be collected from the gingival sulcus.
* After gently drying the area with a blast of air, supragingival plaque will be removed without touching the marginal gingiva. The area will be isolated with cotton rolls to prevent saliva contamination and GCF will be collected by inserting standard paper strips (perio paper; oraflow Inc., Smithtown, NY, USA) into the crevice until mild resistance is felt for 30 seconds.19
* The GCF sample volume will be measured in a calibrated appliance (Periotron 8000 Proflow Inc., Amityville, NY, USA)TM, after which the readings will be converted to an actual volume (µl) by reference to the standard curve. The strips from the selected site will be transferred in micro centrifuged tubes containing 200(µl) of phosphate buffer saline.19

Serum sampling:

* Eight milliliters (8 ml) of blood will be collected from the antecubital fossa after 12 hour fast in the morning using 20-guage needle with 2 ml syringes and will be immediately transferred to the laboratory.
* The blood sample will be allowed to clot at room temperature for one hour, serum will be extracted from blood by centrifuging at 3000 rpm for 15 minutes. Serum sample will be immediately transferred to plastic vial and stored at -800C till the time of assay34 performed using Enzyme Linked ImmunoSorbent Assay (ELISA) kit.

Outcome:

The primary outcome measured will be :

* MMP-8 levels in GCF and serum at baseline and subsequent post surgical follow up after CAF+SCTG procedure (4th ,7th and 6 month).
* Quantitative analysis of GCF samples at baseline and 4th ,7th and 6 month post surgical follow up.
* Correlation of GCF and serum MMP-8 values at baseline and 4th ,7th and 6 month post surgical follow up.

The secondary outcome measured will be :

1. Wound Healing indices (WHI) will be assessed on 4th and 7th day
2. Gingival Recession depth (GRD)
3. Gingival Recession Width (GRW)
4. Probing Depth (PD)
5. Clinical Attachment Level (CAL)
6. Apico coronal width of keratinised tissue (KTW)
7. Plaque Index, Gingival Index and Gingival Bleeding Index

All the above parameters will be correlated with the MMP-8 levels.

Statistical analysis

The values obtained will be compared between the GCF and serum using ANOVA test. Mean differences at different time intervals from the baseline value will be tested using Mann-Whitney U test separately. A 'p' value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* • Miller's Class I and II recession in maxillary anteriors.

  * Patients with thick gingival biotypes >0.8mm.
  * Width of keratinised gingiva >1mm
  * Patients willing to participate in study.
  * Age group of 25-57 years.
  * Patients with history of compliance to oral hygiene instructions and a full mouth plaque score of <20%.(O Leary 1972)
  * American society of Anesthesiologists Physical status I or II.
  * No contra-indications for periodontal surgery.
  * Patients with esthetic concerns.

Exclusion Criteria:

* • Patients with a medical history likely to influence the inflammatory response (atherosclerosis, rheumatoid arthritis, oral cysts, inflammatory bowel disease, bronchiectasis, asthma ,hypertension and diabetes).

  * Recession defects associated with caries/demineralization, restorations, and deep abrasions.
  * No occlusal interferences
  * Teeth with evidence of pulpal pathology.
  * Patients who had received antibiotic therapy within the last 3 months.
  * Pregnant and lactating woman.
  * Patients who have undergone any type of regenerative periodontal therapy six months prior to the initial examination.
  * Patients with history of smoking.
  * Teeth with hopeless prognosis.

Ages: 25 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
MMP-8 levels in GCF and serum and correlation with initial wound healing with recording Wound Healing indices (WHI) assessed on 4th day | subsequent post surgical follow up after CAF+SCTG procedure (4th day post surgery)
MMP-8 levels in GCF and serum and correlation with initial wound healing with recording Wound Healing indices (WHI) assessed on 7th day | subsequent post surgical follow up after CAF+SCTG procedure (7th day post surgery)
Quantitative analysis of GCF samples for mmp-8 in ng/site and its correlation with clinical outcome after 6 months | 6 month post surgical follow up.
Correlation of GCF and serum MMP-8 values | 6 month post surgical follow up

SECONDARY OUTCOMES:
Gingival Recession depth (GRD) | 6 months
Gingival Recession Width (GRW) | 6 months
Apico coronal width of keratinised tissue (KTW) | 6 months
Clinical Attachment Level (CAL) | 6 months
Probing Depth (PD) | 6 months
Plaque Index | 6 months
Gingival Index | 6 months
Gingival Bleeding Index | 6 months